CLINICAL TRIAL: NCT06690502
Title: Safety Profile of Booster IndoVac COVID-19 Vaccination in Healthy Populations Aged 18 Years and Above
Brief Title: Post Authorization Safety Profile of Booster IndoVac COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Other Study IDs: COV19REC-0423
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
Keywords: COVID-19; IndoVac; Safety Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IndoVac COVID-19 Vaccine: Clinically healthy adults aged 18 years and above who received Booster IndoVac COVID-19 Vaccination

SUMMARY:
This study is Post Authorization Safety Study (PASS) Phase IV of Booster IndoVac COVID-19 Vaccination

DETAILED DESCRIPTION:
This study is Post Authorization Safety Study (PASS) Phase IV, to assess any local and systemic reaction after immunization with IndoVac using retrospective cohort study trial design to assess safety profile following IndoVac booster vaccine in healthy populations aged 18 years and above.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy subjects aged 18 years and above
2. Subjects have been injected with IndoVac booster.
3. Minimum 6-month interval from primary or booster COVID-19 vaccination.
4. Subjects have been informed properly regarding the study and signed the informed consent form.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another study when the subjects got IndoVac booster vaccination.
2. Subject's telephone number is invalid or cannot be contacted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 18 years and above
Sampling Method: Non-Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Serious adverse event following IndoVac booster vaccination | until 30 minutes after each dose
  Any serious adverse event occurring from inclusion until 30 minutes after IndoVac booster vaccination

SECONDARY OUTCOMES:
0-7 Days Reactions | Within 0-7 Days after each dose
  Number and percentage of any solicited and unsolicited local reaction and systemic events within 0-7 days after IndoVac booster vaccination.
8-28 Days Reactions | Within 8-28 Days after each dose
  Number and percentage of any solicited and unsolicited local reaction and systemic events within 8-28 days after IndoVac booster vaccination.
28 Days Reactions | 28 Days after each dose
  Number and percentage of any serious adverse event after IndoVac booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hindra Irawan Satari, Prof., Dr., dr., SpA(K), M. Trop. Paed, Principal Investigator — National Committee of Adverse Events Following Immunization / NC Indonesia
Locations (28):
- Indonesia (28):
  - Gambir Public Health Center, Jakarta, Center Jakarta
  - Kemayoran Public Health Center, Jakarta, Center Jakarta
  - Menteng Public Health Center, Jakarta, Center Jakarta
  - Sawah Besar Public Health Center, Jakarta, Center Jakarta
  - Tanah Abang Public Health Center, Jakarta, Center Jakarta
  - Cakung Public Health Center, Jakarta, East Jakarta
  - Cipayung Public Health Center, Jakarta, East Jakarta
  - Ciracas Public Health Center, Jakarta, East Jakarta
  - Makasar Public Health Center, Jakarta, East Jakarta
  - Matraman Public Health Center, Jakarta, East Jakarta
  - Pulogadung Public Health Center, Jakarta, East Jakarta
  - Cilincing Public Health Center, Jakarta, North Jakarta
  - Kelapa Gading Public Health Center, Jakarta, North Jakarta
  - Koja Public Health Center, Jakarta, North Jakarta
  - Pademangan Public Health Center, Jakarta, North Jakarta
  - Cilandak Public Health Center, Jakarta, South Jakarta
  - Jagakarsa Public Health Center, Jakarta, South Jakarta
  - Kebayoran Baru Public Health Center, Jakarta, South Jakarta
  - Mampang Public Health Center, Jakarta, South Jakarta
  - Pancoran Public Health Center, Jakarta, South Jakarta
  - Pesanggrahan Public Health Center, Jakarta, South Jakarta
  - Cengkareng Public Health Center, Jakarta, West Jakarta
  - Grogol Petamburan Public Health Center, Jakarta, West Jakarta
  - Kalideres Public Health Center, Jakarta, West Jakarta
  - Kebon Jeruk Public Health Center, Jakarta, West Jakarta
  - Kembangan Public Health Center, Jakarta, West Jakarta
  - Palmerah Public Health Center, Jakarta, West Jakarta
  - Imunicare Bio Farma, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No